CLINICAL TRIAL: NCT01929239
Title: Phase Ia/Ib Trial of Anti-PSMA Designer T Cells in Prostate Cancer After Non-Myeloablative Conditioning
Brief Title: Trial of Anti-PSMA Designer T Cells in Advanced Prostate Cancer After Non-Myeloablative Conditioning
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-05-1-0408
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Monitor Adverse Events

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti PSMA Designer T Cells (Experimental): Open Label, subjects receive anti PSMA designer T cells, plus IL2, low or moderate dose.
  Interventions: Drug: Anti-PSMA Designer T Cells

INTERVENTIONS:
Drug: Anti-PSMA Designer T Cells

SUMMARY:
This is a Phase Ib Pilot study of anti-PSMA designer T cells in metastatic prostate cancer. Subjects will receive escalating doses of T cells, with either low or moderate dose Interleukin 2. The T cells are collected by pheresis and then genetically modified, and given in a one time infusion.

ELIGIBILITY:
Inclusion Criteria:

5.2.1 Patient with histologically confirmed diagnosis of prostate cancer.

5.2.2 Patient with rising serum PSA,(prostate specific antigen).

5.2.3 Tumor is hormone refractory, as documented by rising PSA with two values separated in time. Patients may enroll if they have a rising PSA after withdrawal of androgen therapy but if enrolled onto this protocol on androgen ablation therapy, they must remain on the androgen therapy for the duration of this protocol. Patients may enroll if tumor is not hormone refractory only if they refuse hormone therapy at this time, and that they understand that hormone therapy is standard treatment for their disease at this stage.

5.2.4 Patient must be at least 18 years of age.

5.2.5 Patient able to understand and sign informed consent.

5.2.6 Patient with a life expectancy of greater than four months.

5.2.7 Patient with performance status of 0 to 1. (http://www.ecog.org/general/perf_stat.html).

5.2.8 Patient with adequate organ function as defined by:

5.2.8.1 ANC 1.0, platelets 50,000, Hgb 8.0; patient may be transfused to achieve Hgb 8.0 to satisfy enrollment criteria, or as otherwise indicated by symptoms for Hgb >8.0.

5.2.8.2 Creatinine 1.5mg/dl or creatinine clearance 60cc/min.

5.2.8.3 Direct bilirubin 1.5 mg/dl.

5.2.8.4 No evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmias, including atrial fibrillation/atrial flutter, evidence of prior myocardial infarction by history or EKG. A normal cardiac stress test for inducible ischemia or arrhythmia within 12 weeks prior to enrollment for all patients over 50 years old or those with abnormal EKG or any history or symptoms suggestive of cardiac disease.

5.2.8.5 No serious, symptomatic obstructive or emphysema¬tous lung disease, or asthma requiring intravenous medications within the past 12 months; no serious lung disease associated with dyspnea at normal activity levels (grade III) or at rest (grade IV), due to any cause (including cancer metastases and pleural effusions). The patient will be ineligible if PFTs show an FEV1 <1.3 liters or a DLCO <50% within 12 weeks of study entry.

For patients enrolling in cohorts IIA, IIB, and III:

5.2.9 Patients with disease in the bone or other site(s) have biopsy-able tumor (at radiologically- or externally-accessible site), and willing to undergo biopsy as specified in 6.3.6. For these groups, patients with >5 lesions bone scan positive lesions will be preferred to increase the yield of blind bone marrow biopsies.

Alternatively, patients with bone or extra-skeletal lesions may be biopsied by CT guided or open procedure.

Exclusion Criteria:

5.3.1 Patients with serious or unstable renal, hepatic, pulmonary, cardiovascular, endocrine, rheumatologic, or allergic disease based on history, physical exam and laboratory tests will be excluded, as outlined in section 5.2.9.

5.3.2 Patients with active clinical disease caused by CMV, hepatitis B or C, HIV or tuberculosis will be excluded from the study.

5.3.3 Patients who have had cytotoxic and/or radiation therapy in the four weeks prior to entry or who have initiated anti-androgen therapy less than six weeks prior to entry will be excluded.

5.3.4 Patients with other concurrent malignancies will be excluded.

5.3.5 Patients requiring systemic steroids will be excluded.

5.3.6 Patients with prior investigational therapies within the 4 weeks prior to entry will be excluded.

5.3.7 Patients previously exposed to mouse antibody will be excluded, unless proven by ELISA to have a negative baseline human anti-mouse antibody (HAMA) titer.

5.3.8 Patients who have had irradiation to whole pelvis or to more than 25% of total marrow will be excluded.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Junghans, PhD, MD, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided